CLINICAL TRIAL: NCT00919412
Title: Non-Invasive Biomarkers To Identify Subjects At Risks For Preterm Delivery
Brief Title: Non Invasive Biomarkers to Identify Subjects at Risk for Preterm Delivery
Acronym: PTMARKER
Status: Terminated | Type: Observational
Why Stopped: Original Principal Investigator, G. Ashmead, MD left the Institution
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 101436-3; 07009
Record Dates: First submitted 2009-06-11; First posted 2009-06-12 (Estimated); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Preterm Birth
Keywords: Non Invasive Biomarkers Preterm Delivery
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Maternal blood Maternal cervical secretions Fetal umbilical cord blood Placenta
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Preterm delivery (< 37 weeks)
- Term delivery (>=37 weeks)

SUMMARY:
The goal of this study is to identify a non-invasive predictor or predictors that will increase the clinician's ability to identify patients with preterm labor (PTL) at risk for preterm delivery (PTD). Through these studies we also hope to reveal potential therapeutic targets in the prevention of prevention of preterm births.

The study hypothesis is that we can identify non-invasive predictors of PTL at risk for PTD.

DETAILED DESCRIPTION:
STUDY DESIGN This is a prospective study involving a cohort of pregnant subjects with pre-term labor. Maternal blood and cervical/vaginal fluid will be collected from consenting subjects with preterm labor. Repeat sampling of cervical fluid will occur as often as weekly until the time of delivery. Relevant clinical and demographic data will be recorded. Levels of prostaglandins (PG's), lipocalin-type prostaglandin D2 synthase (L-PGDS) and cytokines will be determined using ELISA. DNA will also be extracted from maternal blood for SNP analysis of cytokine genes. At the time of delivery, cord blood and placenta samples will be collected if logistically possible (during regular laboratory hours). To determine fetal levels of PG's, L-PGDS and cytokines in cord blood will be analyzed using ELISA. Placental samples will be used for in vitro studies aimed at investigating the placental regulatory pathways of cytokine and PG production. Placental samples will also be processed and embedded in paraffin for use in immunohistochemical studies in order to localize the expression of PG's and cytokines. Clinical delivery data will also be recorded.

Gender of Subjects. Only female subjects will be included.

Age of Subjects. The age of subjects will be restricted to 18-45 years.

Inclusion Criteria. Women with a diagnosis of preterm labor will be included in this study. Preterm labor will be diagnosed as

Six or more contractions per hour associated with one of the following:

1. cervical dilation >= 2 cm
2. cervical effacement > 80%
3. documented changes in dilation or effacement

OR Cervical length less than 2.5 cm by ultrasound with or without contractions.

Exclusion Criteria. Multiple pregnancy, fetal anomalies, abruptio placenta, preeclampsia, cervical dilation greater than 4 cm, clinical signs of infection and vaginal bleeding.

Subject Capacity. All subjects included in this study will have the capacity to give informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Women with a diagnosis of preterm labor.

Exclusion Criteria:

* Multiple pregnancy, fetal anomalies, abruptio placenta, preeclampsia, cervical dilation greater than 4 cm, clinical signs of infection and vaginal bleeding

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women ages 18-45 with a diagnosis of preterm labor
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2007-06; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Preterm delivery | Course of pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Graham G Ashmead, MD, Principal Investigator — Winthrop University Hospital
Locations (1):
- Winthrop-University Hospital, Mineola, New York, United States